CLINICAL TRIAL: NCT04028258
Title: Randomized, Controlled, Crossover, Double-blind Clinical Trial on the Effect of a Mixture of Plant-based Fibers and Carbohydrates on Intestinal Transit in Children Aged 3 to 12 Diagnosed With Functional Constipation
Brief Title: Effect of a Mixture of Fibers and Carbohydrates on Intestinal Transit in Children Diagnosed With Functional Constipation
Acronym: VEGY-DOWN(A)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Ordesa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VEGY-DOWN (A)-05-17
Record Dates: First submitted 2019-07-15; First posted 2019-07-22 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Constipation - Functional
Keywords: Constipation; Fiber
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: study+wash out+control (Other): Study product (3 weeks) + wash out (2 weeks) + control product (3 weeks)
  Interventions: Dietary Supplement: Mixture of fibers + Placebo
- Group B: control+wash out+study (Other): Control product (3 weeks) + wash out (2 weeks) + study product (3 weeks)
  Interventions: Dietary Supplement: Placebo + Mixture of fibers

INTERVENTIONS:
Dietary Supplement: Mixture of fibers + Placebo — Study product: mixture of plant-based food fibers (3 weeks) + wash out (2 weeks) + placebo control : plum flakes + maltodextrin (3 weeks)
  Arms: Group A: study+wash out+control
Dietary Supplement: Placebo + Mixture of fibers — Placebo control: plum flakes + maltodextrin (3 weeks) + wash out (2 weeks) + study product: mixture of plant-based food fibers (3 weeks)
  Arms: Group B: control+wash out+study

SUMMARY:
Once the patients who are candidates to enter the study are identified, the patients will be randomly be assigned to two groups, according to the sequence:

* Group A: study product+wash out+control product
* Group B: control product+wash out+study product

DETAILED DESCRIPTION:
All patients will be given guidelines for adopting dietary habits and healthy lifestyles to achieve a regular and physiological depositional rhythm and will be given a study supplement and a control supplement, alternatively, for 2 time periods of 3 weeks separated by 2 weeks of wash out.

* Supplement under study: mixture of food fibers of plant origin, in a proportion that contributes 75% soluble fiber / 25% insoluble fiber.
* Control: Placebo supplement: maltodextrin and plum flakes

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls aged 3 to 12
* Diagnosis of functional constipation according to Rome IV criteria

Exclusion Criteria:

* Regular use of a dietary fiber supplement, prebiotics or probiotics in the previous 30 days, or who would have been taking bulk-forming agents or laxatives in the 2 weeks prior to the study
* Use of medications that cause constipation
* Children with organic constipation such as Hirschsprung's disease, cerebral paralysis, anorectal and spinal cord abnormalities and metabolic diseases.
* Patients who are not likely to complete follow-up

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of clinical change obtained from the difference between the initial value and the final value for a combined score of the frequency of passage of faeces, pain to defecation, consistency of stool. | From baseline to 8 weeks
  Combined score between this parameters

SECONDARY OUTCOMES:
Consistency of stool according to Bristol Stool Form Scale | From baseline to 8 weeks
  Valuation of stool characteristics (Bristol scale): 7 types of consistency, where type 1 is the hardest consistency.
Frequency of stool | From baseline to 8 weeks
  Equal to or more than 3 times/week, 1-2 times/week, less than 1 time/week
Change in stool weight | From baseline to 8 weeks
  Increase equal to or greater than 50%, increase by 50 - 15%, increase less than 15%
Gastrointestinal symptoms related to the constipation | From baseline to 8 weeks
  Record in the patient's dairy all the gastrointestinal symptoms during the study
Adherence record to the complement intake (Moriski Green test) | At 8 weeks
  4 questions to the patient about treatment adherence.Patients who follow treatment are considered to be those who answer NO to the four questions and not to those who answer YES to one or more.
Patient anthropometric measures: weight | Up to 8 weeks
  Anthropometric records: weight (Kg)
Patient anthropometric measures: size | Up to 8 weeks
  Anthropometric records: size (cm)
Patient anthropometric measures: waist perimeter | Up to 8 weeks
  Waist perimeter (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Rodríguez, MD, Principal Investigator — Instituto de Investigación Sanitaria Aragón
Locations (3):
- Spain (3):
  - Centro de Salud Perpetuo Socorro, Huesca, Aragon
  - Centro de Salud Amparo Poch, Zaragoza, Aragon
  - Centro de Salud Isabel II, Santander, Cantabria